CLINICAL TRIAL: NCT00774215
Title: Retrospective Cohort of the Avaulta Vaginal Mesh Procedure as a Treatment of Pelvic Organ Prolapse
Brief Title: Evaluation of the Avaulta Procedure for the Correction of Pelvic Organ Prolapse - Results at 1 Year
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Patrick Culligan, MD, Director, Division of Urogynecology & Reconstructive Pelvic Surgery, Atlantic Health System
Other Study IDs: R07-09-016
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2008-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Cystocele; Rectocele; Enterocele; Synthetic Mesh; Vaginal Mesh; Transobturator
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Rectocele; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a 1 year review of all patients who had surgery to correct pelvic organ prolapse (i.e. cystocele, rectocele, enterocele) using the Avaulta synthetic mesh kit.

DETAILED DESCRIPTION:
This is a retrospective cohort analysis of all patients who experienced vaginal prolapse and were operated on with the Avaulta synthetic vaginal mesh "kit" from January 2006 to April 2007. The Avaulta synthetic mesh is composed of polypropylene which is a monofilament. The objective of this trial is to compare patients objectively and subjectively at least one year after placement of the Avaulta synthetic vaginal mesh in terms of prolapse symptoms.

This data will be compared to pre-operative data already collected for these patients as a part of their routine surgical work-up. Mesh-related complications will be quantified, including erosions, new-onset pain, and infections. Success and anatomic recurrence rates will be recorded as well

ELIGIBILITY:
Inclusion Criteria:

* All patiAll patients who underwent surgery with the Avaulta synthetic mesh kit from 1/06 - 4/08.

Exclusion Criteria:

* Unable to give informed consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgery with the Avaulta synthetic mesh kit from 1/06 - 4/08.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Anatomical success rates 1 year after surgery to correct pelvic organ prolapse with the Avaulta synthetic mesh kit | 1 year post operatively

SECONDARY OUTCOMES:
Mesh complications 1 year after surgery with the Avaulta synthetic mesh kit | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health System - Division of Urogynecology, Morristown, New Jersey, United States

REFERENCES:
- [Derived] Rudnicki M, Laurikainen E, Pogosean R, Kinne I, Jakobsson U, Teleman P. Anterior colporrhaphy compared with collagen-coated transvaginal mesh for anterior vaginal wall prolapse: a randomised controlled trial. BJOG. 2014 Jan;121(1):102-10; discussion 110-1. doi: 10.1111/1471-0528.12454. Epub 2013 Oct 1. PMID 24118844
- See also: Related Info — http://mybladdermd.com